CLINICAL TRIAL: NCT00063544
Title: Physical Activity and Childhood Obesity
Status: Withdrawn | Type: Observational
Why Stopped: CI left institution
Sponsor: Anna Brooke (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Anna Brooke, Research Governance Officer, University of Bristol
Organization: University of Bristol (Other)
Other Study IDs: 1219; R01HL071248 (NIH)
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To measure associations between physical activity and obesity in a large, population-based cohort of children.

DETAILED DESCRIPTION:
BACKGROUND:

Childhood obesity is rapidly increasing in many countries and environmental factors are the main cause. The onset of puberty may be a critical period. Diet and physical activity are likely to be prime causative factors, although the relative role of each may vary between children of differing age, gender and ethnicity. There are also likely to be many psychosocial and social-demographic factors that can confound these relationships, and these confounders may vary between sub-groups. There continues to be uncertainty regarding the role of these factors and their differential effects in subgroups of the population. It is crucial to develop a better understanding of how dietary and physical activity patterns affect energy balance, and how these characteristics interact with other factors.

Measures of physical activity will be added to ongoing assessments of boys and girls (n=10,000) participating in the Avon Longitudinal Study of Parents and Children (ALSPAC). This comprehensive study has been following children and their parents for about 9-10 years. The study has an extensive database including maternal and paternal social background, lifestyle and habits (including diet and physical activity), medical history and medications during pregnancy and thereafter. ALSPAC has also collected and retained biological samples including maternal blood, urine, cord blood, umbilical cord, placenta, hair and nail clippings, deciduous teeth, child's blood and DNA. Data on the mothers also include details of her own parent's lifestyle, her childhood, lifestyle, occupation history and diet, and access to mother's biological samples. Over 71% of the cohort (>10,000 of 14,541 participants) have been retained.

DESIGN NARRATIVE:

Levels and patterns of physical activity will be measured on all children at ages 11 and 13 to assess relationships with measures of obesity. Physical activity will be measured objectively for 5 days. The data, together with other data collected during pregnancy, infancy and childhood will be used to investigate relationships between modes, intensities, quantities and patterns of physical activity and the development of obesity at this critical stage of life. The strengths of this prospective study are its size, high retention rates and the extensive set of whole-of-life measures already taken on the children. With over 10,000 children expected to attend annually for health checks throughout adolescence, the study will be adequately powered to quantify associations between physical activity and obesity. The study of physical activity in children has to date been seriously restricted because of high levels of measurement error inherent in all self-report measures of physical activity. In this study, physical activity will be measured using a single-plane accelerometer (CSA model 7164) - a small, lightweight electronic motion sensor attached to the child's belt for a period of 5 days. This instrument gives the capacity to to characterize children's physical activity, and inactivity, more accurately than ever before. Comprehensive measurements of diet and body composition (principally Dual-emission X-ray Absorptiometry - DXA) will also be taken at ages 11 and 13 under separate funding.

ELIGIBILITY:
No eligibility criteria - Not an applicable clinical trial

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Not an applicable clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Levels and patterns of physical activity will be measured on all children at ages 11 and 13 to assess relationships with measures of obesity. | 5 days
  In this study, physical activity will be measured using a single-plane accelerometer (CSA model 7164) - a small, lightweight electronic motion sensor attached to the child's belt for a period of 5 days. This instrument gives the capacity to to characterize children's physical activity, and inactivity, more accurately than ever before.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Riddoch, Principal Investigator — Bristol University